CLINICAL TRIAL: NCT02055027
Title: Adherence to Continuous Positive Airway Pressure Among Obstructive Sleep Apnoea Patients. An Anaesthetic Algorithmic Approach to Prevent Postoperative Complications.
Brief Title: Adherence to Continuous Positive Airway Pressure Among Obstructive Sleep Apnoea Patients.
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Eric DEFLANDRE, MD, FCCP, Astes
Other Study IDs: ASTES-NCPAP
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep Apnea, Obstructive; Continuous Positive Airway Pressure; Perioperative Period
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adherent Patients: Comparison between groups
  Interventions: Other: Comparison between groups
- Non-adherent patients: Comparison between groups
  Interventions: Other: Comparison between groups

INTERVENTIONS:
Other: Comparison between groups — Comparison between the two groups (adherent and non-adherent patients) in order to discover criteria of non-adherence

SUMMARY:
Prospective study designed to identify factors that would predict patient adherence to CPAP (Continuous Positive Airway Pressure) therapy.

DETAILED DESCRIPTION:
Prospective study designed to identify factors that would predict patient adherence to CPAP therapy.

Comparison between data recorded among patients and the data of the CPAP microchip.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 patients)
* All patients under CPAP (Continuous Positive Airway Pressure) therapy coming for annual visit in the Sart-Tilman Sleep Study Center

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sleep Study Center
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Number of hours of CPAP use by night | Baseline
  Analyse of the data recorded by the CPAP microchip in order to assess the adherent or non-adherent status to the patient (adherent: CPAP use > 4 hours per night, non-adherent: less than 4 hours)

SECONDARY OUTCOMES:
Lickert's scale to assess criteria of non-adherence | Baseline
  Evaluation of 72 criteria by a Lickert's scale in order to assess characteristics associated with non-adherence to CPAP therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Centre Hospitalier Universitaire (CHU) Sart-Tilman, Liège, Liege, Belgium